CLINICAL TRIAL: NCT06416904
Title: Evaluation Of Anchorage Control Using Arch Wire Stopper in Comparison to Mini-Screws in Post-Pubertal Patients: A Randomized Clinical Trial
Brief Title: Evaluation Of Anchorage Control Using Arch Wire Stopper Versus Mini-Screws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennatallah Moamen Mohamed Mohamed Ali, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTH3-3-3
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arch wire stopper mesial to the maxillary first molar group (Experimental): In postpubertal female patients with maxillary dentoalveolar protrusion, canine retraction after the extraction of the maxillary first premolars with archwire stoppers mesial to the maxillary first molars followed by anterior segment retraction using T-loop on 0.017x0.025 TMA arch wire.
  Interventions: Device: archwire stopper mesial to the maxillary first molar group
- maxillary first molar indirectly anchored to the inter-radicular mini-screw group (Active Comparator): In postpubertal female patients with maxillary dentoalveolar protrusion, canine retraction after the extraction of the maxillary first premolars, with the maxillary first molars indirectly anchored to the inter-radicular mini-screw followed by anterior segment retraction using T-loop on 0.017x0.025 TMA arch wire.
  Interventions: Device: inter-radicular mini-screw

INTERVENTIONS:
Device: archwire stopper mesial to the maxillary first molar group — canine retraction after the extraction of the maxillary first premolars with archwire stoppers is mesial to the maxillary first molars.
  Arms: arch wire stopper mesial to the maxillary first molar group
Device: inter-radicular mini-screw — canine retraction after the extraction of the maxillary first premolars, with the maxillary first molars indirectly anchored to the inter-radicular mini-screw.
  Arms: maxillary first molar indirectly anchored to the inter-radicular mini-screw group

SUMMARY:
The study aims to compare the anchorage control using arch wire stopper versus mini-screws in post-pubertal patients with maxillary dentoalveolar protrusion

DETAILED DESCRIPTION:
The study begins with patient selection according to inclusion and exclusion criteria, followed by treatment planning, and then bonding of orthodontic brackets of the upper and lower arches, including the second maxillary molars.

After leveling and alignment for all participants, the extraction of the maxillary first premolars will be performed.

• In the "Intervention Group" Canine retraction will be performed on 0.017×0.025 ss archwire with an archwire stopper mesial to the upper first molar.

Afterwards, anterior segment retraction will be done using T-loop on 0.017x0.025 TMA archwire

• In the "Comparator Group" Canine retraction on 0.017×0.025 ss archwire with the upper first molars indirectly anchored to inter-radicular mini screws Afterwards, anterior segment retraction will be done using T-loop on 0.017x0.025 TMA archwire

Lastly, the anchorage control in both groups and the secondary outcomes will be assessed using the obtained digital models and lateral cephalometric radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Post-pubertal female patients.
* Cases with bimaxillary protrusion or Class II Division 1 malocclusion that require maxillary first premolars extraction.
* Full permanent dentition (not necessitating third molars).
* Good oral hygiene.

Exclusion Criteria:

* Medically compromised patients.
* Active periodontal disease or obvious bone loss in the maxillary arch.
* Patients with habits that are detrimental to dental occlusion (thumb sucking, tongue thrusting).
* Smoking or any systemic diseases.
* Chronic use of any medications including antibiotics, phenytoin, cyclosporine, anti-inflammatory drugs, systemic corticosteroids, and calcium channel blockers. All the above factors affect the rate of tooth movement
* Previous orthodontic treatment.
* Missing teeth.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — female patients 15-25 years
Enrollment: 26 (Actual)
Dates: Start 2024-02-13 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Amount of anchorage loss of the maxillary first molars | 6 months from the start of the canine retraction and after anterior segment retraction (12 months)
  After full canine retraction, the amount of anchorage loss (mesial movement) of the maxillary first molars of will be assessed on the digital models

SECONDARY OUTCOMES:
Tipping of the maxillary first molar. | 6 months from the start of the canine retraction and after anterior segment retraction (12 months)
  the degree of tipping of the maxillary first molars will be assessed on the lateral cephalometric radiograph
Maxillary incisors inclination | 6 months from the start of the canine retraction and after anterior segment retraction (12 months)
  The change in the maxillary incisors inclination will be assessed on the lateral cephalometric radiograph
Maxillary incisors anteroposterior position | 6 months from the start of the canine retraction and after anterior segment retraction (12 months)
  The change in the maxillary incisors anteroposterior position will be assessed on the lateral cephalometric radiograph and digital models

CONTACTS AND LOCATIONS:
Overall Officials: Mennatallah Ali, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No